CLINICAL TRIAL: NCT06216379
Title: Is Sensory Processing Associated With Gross and Fine Motor Skills at 1-Year-Old?
Brief Title: Sensory Processing Associated With Motor Skills
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Gazi University, Gazi University
Other Study IDs: E-77082166-604.01.02-739050
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth; Sensory Processing Disorder; Motor Delay
MeSH Terms: conditions — Premature Birth; Psychomotor Disorders | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm: Children born before 37 gestational weeks
  Interventions: Diagnostic Test: Assessment
- Term: Children born after 37 weeks of gestation
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — Sensory processing skills and gross and fine motor development of preterm and term born children were evaluated.

SUMMARY:
In the study, sensory processing skills of 1-year-old preterm and term children will be evaluated. The relationship between sensory processing skills and gross and fine motor development will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Premature group: Healthy children with a gestational age below 34 weeks Term group: Healthy children with gestational age between 37-41 weeks

Exclusion Criteria:

they had major congenital malformations, had genetic or chromosomal abnormalities, had known metabolic disorders, or had seizures.

Ages: 12 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: Healthy children born preterm and term at 12 months of age
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Test of Sensory Functions in Infants TSFI | 15 minutes
  The Test of Sensory Functions in Infants (TSFI) is a standardized and reliable tool designed to evaluate the sensory development of infants aged 4-18 months. Consisting of 24 items, the TSFI measures reactions in five distinct subdomains: tactile deep pressure, visual-tactile integration, adaptive motor function, ocular motor function, and reactivity to vestibular stimulation [1]. A specific age-normalized score is generated for each subdomain, contributing to a total score determined by the sum of all subdomains. The total score ranges from 0 to 49, with higher scores indicating more typical sensory responsiveness and lower scores suggesting behaviors associated with sensory over-responsivity [2]. In this study, a physiotherapist administered the TSFI to assess the sensory development of infants.

SECONDARY OUTCOMES:
Peabody Developmental Motor Scales-2 | 30 minutes
  The PDMS-2 is a widely employed and acknowledged assessment tool for evaluating a child's motor abilities. Its primary purpose is to distinguish and aid in identifying developmental delays in children aged 5 and below by comparing their performance against established norms [3]. The gross motor skills section includes 4 subtests: reflexes, stationary, locomotion, and object manipulation. Similarly, the fine motor skills segment consists of 2 subtests: grasping and visual-motor integration. Each item in the test is evaluated using a 3-point scoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)